CLINICAL TRIAL: NCT07186218
Title: Use of an Electronic Patient-Reported Outcome Measure for Symptom Monitoring With Supported Feedback in Advanced Chronic Kidney Disease
Brief Title: Symptom Monitoring With Supported Feedback in Advanced Chronic Kidney Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Kendra Wulczyn, MD, Physician, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024p002276; 1K23DK140642-01A1 (NIH)
Record Dates: First submitted 2025-09-10; First posted 2025-09-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Disease (Stages 4 and 5); Health Related Quality of Life
Keywords: chronic kidney disease; health related quality of life; patient-reported outcome measure; chronic kidney disease associated symptoms
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: The design is a single-center, open-label, randomized pilot trial examining the implementation and preliminary efficacy of an electronic PROM (ePROM) for routine symptom assessment with feedback of responses to clinicians among adults living with advanced CKD (eGFR <30 mL/min/1.73m2). Patients will be assigned to either the ePROM group (35 patients) or the Usual Care group (35 patients).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic patient-reported outcome (ePROM) intervention for routine symptom assessment (Active Comparator): The ePROM intervention consists of: 1) Patient reporting of CKD-related symptoms at regular intervals using an electronic version of the Integrated Patient Outcome Scale (IPOS)-Renal survey; 2) Feedback of patient responses to clinicians, and 3) Provision of guidance for symptom management to clinicians. Patients randomized to the ePROM intervention will be asked to complete monthly reporting of CKD-associated symptoms.
  Interventions: Behavioral: Electronic patient-reported outcome measure (ePROM) for symptom monitoring
- Usual Care (No Intervention): For patients randomized to Usual Care, there will be no study-driven changes to existing clinical practices for patient symptom reporting or clinician follow-up of patient-reported symptoms. Usual care symptom monitoring consists of patients and clinicians discussing symptoms at their own discretion. Under usual care, no symptom guidance documents or patient symptom reports are provided to clinicians.

INTERVENTIONS:
Behavioral: Electronic patient-reported outcome measure (ePROM) for symptom monitoring — Patients randomized to the ePROM intervention arm will be asked to complete monthly reporting of their CKD-associated symptoms using an electronic version of the Integrated Patient Outcome Scale (IPOS)-Renal survey. Their responses will be provided in summary form to their nephrology clinicians at regular intervals and prior to any nephrology clinic visits. Clinicians will be provided with guidance on symptom management and will have the option to participate in an informational session on how to interpret patient symptom responses.
  Arms: Electronic patient-reported outcome (ePROM) intervention for routine symptom assessment

SUMMARY:
Patient-reported outcome measures (PROMs) are validated tools to reliably measure outcomes highly prioritized by patients, such as health-related quality of life (HRQOL) and symptoms, but the current clinical impact of PROMs is limited by a lack of evidence-based methods to incorporate them into routine care. Symptoms, which are highly prevalent among persons living with chronic kidney disease (CKD), substantially contribute to the reduced HRQOL experienced by this patient population. HRQOL spans several domains of wellbeing affected by disease, including physical, mental, and social health, functionality, and symptoms. Both HRQOL and symptom burden are consistently identified by patients with CKD as top clinical and research priorities. These issues are particularly salient to individuals living with advanced CKD, who suffer significant symptom burden that is often underrecognized and undertreated by nephrology providers, yet is a key factor considered by nephrologists for the timing of dialysis initiation. Randomized controlled trials of patients with other chronic illnesses show that routine assessment of symptoms with PROMs improves symptom burden, patient-provider communication, and HRQOL; yet, standardized approaches to regular symptom monitoring among patients with advanced CKD are lacking. This pilot, randomized trial of a PROM-based intervention for routine symptom reporting by patients with feedback of responses to nephrologists aims to address the lack of data on PROM use for symptom assessment in nephrology care. We will evaluate the implementation (reach, feasibility, and acceptability) and preliminary efficacy of monthly patient report of CKD-related symptoms using the electronic IPOS-Renal questionnaire with supported clinician follow-up for 12 months versus standard of care. This trial will utilize complementary quantitative and qualitative methods to evaluate the implementation of the PROM-based intervention. The results of this pilot study will inform a definitive, cluster-randomized trial on the effect of a PROM-based symptom assessment intervention to improve HRQOL and clinical outcomes among patients living with advanced CKD.

DETAILED DESCRIPTION:
This is a single-center, open-label, two-arm, randomized pilot trial of 70 individuals with advanced chronic kidney disease (CKD; eGFR<20 mL/min/1.73 m2). This pilot study will assess reach, feasibility, acceptability (implementation) and preliminary efficacy of patient use of IPOS-Renal (Integrated Patient Outcome Scale-Renal, primary exposure of interest), an instrument designed to assess symptoms among patients with CKD, which will be electronically completed monthly for 12 months. Randomization will occur in a 1:1 ratio at the level of the individual; therefore, 35 individuals will be randomized to the IPOS-Renal electronic patient-reported outcome measure (ePROM) intervention arm, and 35 individuals will be randomized to the control arm (standard of care).

The ePROM intervention has three core components: 1) patient self-reporting of CKD-related symptoms at regular intervals using the Integrated Patient Outcome Scale (IPOS)-Renal survey, 2) feedback of patient responses to clinicians; and 3) provision of guidance for symptom management to clinicians. Patients randomized to the ePROM intervention arm will receive instruction on how to self-report symptoms using an electronic version of the IPOS-Renal instrument. Clinicians will be provided instruction on how to view patient symptom responses and given guidance regarding symptom management strategies; however, treatment decisions will be left entirely to the discretion of the clinician. Whenever a patient has a clinic visit, a symptom report will be generated and printed by the research team and will be given to the treating nephrologist.

All participants will complete two PROMs over the course of participation. At baseline, participants will complete the Kidney Disease Quality of Life-36 (KDQOL) instrument (primary efficacy outcome) and the IPOS-Renal to assess symptom burden at baseline. Participants will be given a choice to complete questionnaires online, via mailed paper forms, or over the telephone. The KDQOL questionnaire will be completed at baseline and months 6 and 12 (+/- 4 weeks each). All study questionnaires will be available in English. Chart abstraction will be conducted by a member of the study team at baseline, 3, 6, 9, and 12 months (+/- 1 months each) to collect demographic and clinical data. Additional information on clinical events (progression to CKD requiring kidney replacement therapy, emergency room visits, hospitalizations, and death) will be abstracted at 24 months. Patient and clinician participants (target n=20 patients and n=10 clinicians) will be invited to participate in semi-structured interviews for qualitative data collection. Qualitative data will be used to explore patient and clinician perspectives on symptom management in the ambulatory nephrology setting and the feasibility and acceptability of the ePROM intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years)
* Advanced CKD, defined as at least two measurements of creatinine-based or cystatin C-based eGFR ≤ 30 mL/min/1.73m2 separated by at least 90 days in the preceding 12 months
* Able to provide consent to participate in the study
* Able to read and write in English
* Under the care of a nephrologist at a Mass General Brigham nephrology clinic

Exclusion Criteria:

* Terminal illness likely to lead to death within 6 months of participation
* Patients receiving dialysis treatment at the time of enrollment or scheduled to start dialysis therapy in the next 4 weeks
* Patients scheduled to receive a kidney transplant in the next 6 months
* Patients having their initial clinic visit (i.e., new to the clinic)
* Cognitive deficits that would preclude understanding of consent form and/or questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Reach (Implementation); Screen-eligibility | Baseline
  Percent of screen-eligible patients from pool of patients with advanced CKD screened for eligibility.
Reach (Implementation); Rate of consenting | Baseline
  Percent of screen-eligible patients approached to participate in study who provide consent to participate
Feasibility (Implementation); symptom survey completion rate | Duration of active 12-month study participation
  Rate of completion of electronic symptom questionnaires by participants
Feasibility (Implementation); Symptom documentation | Duration of active 12-month study participation
  Frequency of symptom documentation by clinicians in the clinical visit note for participants
Feasibility (Implementation); Interviews | 3-12 months of participation
  Clinician and patient participant answers to interview questions regarding the extent to which the ePROM intervention fits within the ambulatory nephrology setting.
Acceptability (Implementation); Interviews | 3-12 months of participation
  Clinician and patient participant answers to interview questions regarding satisfaction with and acceptability of the ePROM intervention.

SECONDARY OUTCOMES:
Progression to End-Stage Kidney Disease | Duration of active 12-month study participation plus 12 months; 24 months total
  Rate of progression to end-stage kidney disease requiring kidney replacement therapy (i.e., initiation of dialysis treatment or receipt of a preemptive kidney transplant)
Emergency Room Visits | Duration of active 12-month study participation plus 12 months; 24 months total
  Rate of visits to the Emergency Room
Hospitalizations | Duration of active 12-month study participation plus 12 months; 24 months total
  Hospitalization rate
Mortality | Duration of active 12-month study participation plus 12 months; 24 months total
  Mortality rate

OTHER OUTCOMES:
Health-Related Quality of Life: Kidney Summary Score (Preliminary Efficacy) | Baseline, 6 months, 12 months
  Kidney Disease Quality of Life-36 (KDQOL-36) This outcome will be assessed as change in the kidney summary score of the KDQOL-36 over 12 months. Lowest score - 0; Highest score - 100. A lower score indicates a worse outcome.
Health-related quality of life: Physical (Preliminary Efficacy) | Baseline, 6 months, 12 months
  Kidney Disease Quality of Life-36 (KDQOL-36)
  This outcome will be assessed as change in the physical composite score of the KDQOL-36 over 12 months. Lowest score - 0; Highest score - 100. A lower score indicates a worse outcome.
Health-Related Quality of Life: Mental (Preliminary Efficacy) | Baseline, 6 months, 12 months
  Kidney Disease Quality of Life-36 (KDQOL-36) This outcome will be assessed as change in the mental composite score of the KDQOL-36 over 12 months. Lowest score - 0; Highest score - 100. A lower score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No